CLINICAL TRIAL: NCT01081938
Title: National, Phase IV, Multicentric, Open Label, Comparative Study to Evaluate the Efficacy and Safety of Insulin Glargine Plus Glulisine and Sliding Scale Plus Glulisine in Hospitalized Patients With Diabetes Metabolism Type II Under Enteral Nutrition.
Brief Title: Insulin Glargine for Diabetes Metabolism(DM)Type II Patients Under Enteral Nutrition
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_04572; U1111-1116-9777 (Other: UTN)
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Insulin Glargine + Insulin Glulisine
  Interventions: Drug: INSULIN GLARGINE; Drug: INSULIN GLULISINE
- 2 (Active Comparator): Insulin Glulisine
  Interventions: Drug: INSULIN GLULISINE

INTERVENTIONS:
Drug: INSULIN GLARGINE — Pharmaceutical form: Lantus® (100 U/ml)
  Route of administration: Subcutaneous injection with SoloStar® (3 ml) pen device.
  Dose regimen: Single daily dose of Insulin Glargine
  Arms: 1
Drug: INSULIN GLULISINE — Pharmaceutical form: Apidra® (100 U/ml)
  Route of administration: Subcutaneous injection with SoloStar® (3 ml) pen device
  Dose regimen:
  Arm1: Every 6 hours Arm2: several daily dose according to sliding scale of Insulin Glargine

SUMMARY:
Primary Objective:

1- Proportion of patients with mean daily glycemia <140mg/dL during the period of 7 days of treatment with glargine plus supplemental glulisine versus patients with glulisine sliding scale.

Secondary Objective:

1. Incidence of moderate hyperglycemia (>140mg/dL) during the treatment period.
2. Incidence of hypoglycemia (<60mg/dL and < 40mg/dL) during the treatment period.
3. Incidence of severe hyperglycemia (>400mg/dL) during the treatment period.
4. Total dose of insulin and correction dose in each group.

ELIGIBILITY:
Inclusion criteria:

* Men and women with type 2 diabetes that will need enteral nutrition with carbohydrate content.
* Glycemia >140mg/dL and < 400mg/dL at admission on the ward.
* Informed consent (patient or legally authorized representative)

Exclusion criteria:

* Hypersensibility to insulin glargine or glulisine, or any other component of the insulin formulation.
* Use of investigational medications during the last 12 months or use of any investigational insulin preparation during the last 4 months.
* History of diabetic ketoacidosis or hyperosmolar hyperglycaemic state or ketonuria.
* Subjects with conditions that are expected to need surgery or intensive care unit (ICU)admission based on discussions with the treatment team and attending physician.
* Pregnancy.
* Severe hepatic disease or active hepatitis.
* Cardiac failure class III or IV (Classification de la New York Heart Association:NYHA).
* Diagnosed advanced autonomic neuropathy.
* Diagnosed cancer.
* Active infection.
* Current therapy with steroids.
* Patients with recognized or suspected endocrine disorders associated with increased insulin resistance, acromegaly, or hyperthyroidism.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Glycaemic parameters assessment | During the period of 7 Days of treatment

SECONDARY OUTCOMES:
Incidence of moderate and severe hyperglycemia | During the period of 7 Days of treatment
Incidence of symptomatic, nocturnal and severe hypoglycemias | During the period of 7 Days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- Brazil (10):
  - Sanofi-Aventis Investigational Site Number 076-007, Belo Horizonte
  - Sanofi-Aventis Investigational Site Number 076-011, Curitiba
  - Sanofi-Aventis Investigational Site Number 076-005, Joinville
  - Sanofi-Aventis Investigational Site Number 076-001, Porto Alegre
  - Sanofi-Aventis Investigational Site Number 076-004, Porto Alegre
  - Sanofi-Aventis Investigational Site Number 076-006, São José do Rio Preto
  - Sanofi-Aventis Investigational Site Number 076-010, São Paulo
  - Sanofi-Aventis Investigational Site Number 076-008, São Paulo
  - Sanofi-Aventis Investigational Site Number 076-003, São Paulo
  - Sanofi-Aventis Investigational Site Number 076-009, São Paulo